CLINICAL TRIAL: NCT07247565
Title: Comparative Study Between Conventional Radiofrequency Ablation vs Chemical Neurolysis of Ganglion Impar for Treatment of Chronic Non Cancer Related Coccydynia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lydia edward aziz zakhary, lecturer of anesthesia , intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: non cancer coccydynia
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pain Management
Keywords: coccydinea; pain; radiofrequency; alcohol neurolysis
MeSH Terms: conditions — Agnosia; Pain | interventions — Radiofrequency Ablation; Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- radiofrequency group (Active Comparator): patients with non cancer coccydynia in this group will receive conventional radiofrequency on ganglion impar
  Interventions: Procedure: Radiofrequency ablation alone
- alcohol neurolysis group (Experimental): patients in this group will receive alcohol neurolysis on ganglion impar
  Interventions: Procedure: Alcohol injection

INTERVENTIONS:
Procedure: Radiofrequency ablation alone — The entry site was detected under fluoroscopy then local anesthesia was given using lidocaine 2% followed by the insertion of a radiofrequency cannulas (STRYKER 20 G, 9 cm with 1 cm active tip) targeting the junction between the coccygeal bones and pass through it anteriorly in the lateral view. Finally confirming the proper site with a contrast dye in lateral and A-P views.
  10 ml of lidocaine 1 % was injected to tolerate the ablation then in the 1st group placing of the radiofrequency cable followed by ablation will be done at 80 degrees for 90 seconds.
  Arms: radiofrequency group
Procedure: Alcohol injection — The entry site was detected under fluoroscopy then local anesthesia was given using lidocaine 2% followed by the insertion 22 G spinal needle targeting the junction between the coccygeal bones and pass through it anteriorly in the lateral view. Finally confirming the proper site with a contrast dye in lateral and A-P views.
  10 ml of lidocaine 1 % was injected to tolerate the ablation then injection of 5 ml 70% alcohol will be performed
  Arms: alcohol neurolysis group

SUMMARY:
Aim: compare effectiveness (satisfaction) and duration of pain relief between patients who perform the conventional thermal radiofrequency on the ganglion impar vs patients who perform the chemical neurolysis with alcohol in patients with non cancer coccydynia patients with non cancer coccydynia not responding to medical treatment will be divided into 2 groups before intervention , control group will receive conventional radiofrequency ablation of ganglion impar , while the study group will receive alcohol neurolysis

ELIGIBILITY:
Inclusion Criteria:

* non cancer coccydynia

  1. Both genders
  2. Age between 20-70 years.
  3. ASA 1,2 & 3 physical status
  4. xray coccyx lateral position showing normal joints and bones with no fractures

Exclusion Criteria:

* Neurological disorders. (previous central and peripheral CNS affection).

  * coagulopathy INR > 1.8 or platelets < 50,000.
  * Infection at or near the injection site.
  * Presence of pacemaker or defibrillator.
  * known allergy to used medications.
  * patients with previous history of Radiotherapy, chemotherapy or metastasis
  * pregnant patients.
  * patients with rheumatological disorders (rheumatoid arthritis, diffuse idiopathic skeletal hyerostosis, psoriatic arthritis)
  * age <20 or >70
  * Xray coccyx showing fractures or abnormalities

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
pain relief using Numeric Pain score scale | 1 month
  patients will be asked to describe their pain on Numeric pain scale ( an 11 numbers scale where 0 describes no pain and 10 describes the worst pain ) and compare it to before the procedure
pain relief of chronic non cancer coccydynia | 6 months after the procedure
  patients will be asked to describe their pain on Numeric pain scale and compare it to before the procedure
patient global impression of change (PGIC) | 6 months
  one-item questionnaire that asks patients to rate their overall improvement after a treatment.he scale typically includes ratings such as "very much improved," "much improved," "minimally improved," "unchanged," or "worse".

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fogel GR, Cunningham PY 3rd, Esses SI. Coccygodynia: evaluation and management. J Am Acad Orthop Surg. 2004 Jan-Feb;12(1):49-54. doi: 10.5435/00124635-200401000-00007. PMID 14753797